CLINICAL TRIAL: NCT02009566
Title: Healthy Volunteer Visibility Study of Micromachined Tags for the Detection of Surgical Sponges
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Initial PI Dr. Marentis left the University of Michigan hospital
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Aine Kelly, MD, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM00063233
Record Dates: First submitted 2013-11-11; First posted 2013-12-12 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Injury Due to Foreign Object Accidentally Left in Body During Surgical Operation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abdominal radiographs with microfabricated tags (Experimental)
  Interventions: Radiation: Abdominal radiographs with microfabricated tags

INTERVENTIONS:
Radiation: Abdominal radiographs with microfabricated tags — Subjects will have 2 x-rays of their lower thorax/ abdomen taken. For each x-ray, a microfabricated tag or no tag will be placed in a different position. The x-rays will take approximately 15 minutes to complete.
  Other Names: Abdominal CT (computerized tomography)

SUMMARY:
Surgical sponges can be accidentally left inside patient's bodies. We are working on special tags (called microfabricated tags) that surgeons can put on their sponges. Then, if the surgeons forget to remove a sponge from a patient, they'll be able to detect these special tags in an x-ray.

DETAILED DESCRIPTION:
Surgical sponges can be accidentally left inside patient's bodies. We are working on special tags (called microfabricated tags) that surgeons can put on their sponges. Then, if the surgeons forget to remove a sponge from a patient, they'll be able to detect these special tags in an x-ray. We wish to take x-rays of healthy people's abdomens with microfabricated tags lying on them. The x-rays will help us improve our system for detecting sponges left inside people's bodies.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women
2. Ages 18 or older -

Exclusion Criteria:

1. Under 18 years of age
2. Pregnant female or if female has not had a negative pregnancy test prior to the research scans.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Validate the CAD (computer aided detection) system | 3 years
  X-rays of the microfabricated tag will be taken. These x-rays will be reviewed and the individual tags identified manually and a control file created. The images will then be processed by the CAD (computer aided detection)system and the output will be compared to the control file.

CONTACTS AND LOCATIONS:
Overall Officials: Aine Kelly, MD, Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No